CLINICAL TRIAL: NCT05997407
Title: The Effect of a Mindset Management Approach on Stress Levels in Women With Infertility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Shady Grove Fertility Reproductive Science Center (Other)
Responsible Party: Principal Investigator, Emily Evans-Hoeker, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB # 23-241
Record Dates: First submitted 2023-07-26; First posted 2023-08-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Stress; Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Organic Conceptions intervention group (Experimental): Will complete Organic Conceptions intervention.
  Interventions: Behavioral: Organic Conceptions mindset management program
- Control group (No Intervention): Will not complete Organic Conceptions intervention.

INTERVENTIONS:
Behavioral: Organic Conceptions mindset management program — Organic Conceptions is a theoretical model and corresponding 9-step cognitive-based therapy program that enables people to understand where they are in their fertility journey, and provides them with coping strategies to reframe the painful emotional side effects of infertility. In addition to the 9-step program, there are mini-classes on the key triggers that people face when dealing with infertility.
  The intervention consists of a series of assignments that participants in the intervention group will complete for a ten-week period. These assignments will take approximately three hours per week to complete. In addition, participants will complete biweekly live support group sessions led by certified coaches and will have the option to join a Facebook support group.
  Arms: Organic Conceptions intervention group

SUMMARY:
The goal of this clinical trial is to test the effect of a mindset management intervention on stress levels in women with infertility. The main question it aims to answer is:

Can the Organic Conceptions approach decrease stress levels in women with infertility?

Participants in both groups will be asked to complete three surveys at three time points. The intervention group will complete the Organic Conceptions program, while the control group will not complete an intervention.

Researchers will compare the intervention group and control group to see if the Organic Conceptions mindset management program decreases stress levels in women with infertility.

DETAILED DESCRIPTION:
The study follows a randomized controlled, unblinded, between-groups, and repeated measure design. The study period will last 16 weeks for both groups. Potential subjects will first be screened by a patient service representative at the SGF office in Roanoke, who will generate a report of new patients who were seen recently. The patient service representative will then reach out to those patients via email and introduce them to the study. If they are interested in enrolling, they will fill out the REDCap survey linked in the email, which asks for their name, email, and phone #. If they fill out the survey, a designated study team member will call them and verify the patient by name. Designated study team members include clinical research personnel at SGF, co-investigators at Virginia Tech, the Principal Investigator, and medical students at Virginia Tech. The designated study team member will introduce the patient to the study. If they are interested in enrolling, they will confirm their eligibility, and review the consent form with the patient. Participants will sign the eConsent using a finger or mouse to sign. The participants will sign the consent form while having a conversation over the phone with a designated study team member. The designated study team member will verify that the participant's signature has been saved correctly in REDCap. If participants don't answer their phone, the designated study team member may email them to set up a time to discuss the study. Participants will be randomized to one of two groups: the OC research-related intervention group or the control group. Participants will then be sent instructions on next steps, based on their randomization result.

Throughout the study period, subjects will complete surveys through REDCap. These will be emailed to them. Surveys will include a demographics questionnaire, the COMPI-FPSS, the Client Satisfaction Questionnaire for Internet Interventions CSQ-I, and additional questions. Demographic questionnaire components were developed based on previous research (Clifton et. al 2020, Kirca et. al 2019) and include questions on age, gender, relationship status, length of current relationship, number of pregnancies, number of living children, ethnicity, race, income, employment status, highest level of education, type of area patient resides in, mental conditions, and current use of therapeutic interventions. The COMPI-FPSS is a measure of fertility-related stress (Sobral et. al 2016). It is based on the Fertility Problem Inventory (FPI) (Abbey et. al 1991) and an interview study completed in couples, which analyzed the psychosocial consequences of infertility (Schmidt et. al 2006). The scale is a reliable and validated measure of stress, specifically related to infertility, that can be applied in various cultures and countries (Sobral et. al 2016). Compared to two other known infertility-specific psychometric measures (FPI and Fertility Quality of Life), the COMPI-FPSS has a practical advantage due to its shorter length, and it differentiates most effectively between its domains (Pedro et. al 2016), which include a personal, marriage, and social domain. With the permission of Dr. Schmidt, the creator of the COMPI-FPSS, the marriage domain is labeled a "relationship" domain in order to encompass all types of relationships. If the patient is not in a relationship, then the relationship domain questions will be omitted. The COMPI-FPSS includes questions about infertility-related stress, specifically, rather than general stress. This makes it a reliable tool because it controls for stress from other aspects of life. It employs a Likert scale, which includes a variety of statements that participants may choose from when responding to qualitative questions. Participant scores will be added and analyzed within each domain and overall. A higher score means higher stress levels, while a lower score means lower stress levels. The CSQ-I is a reliable measure for Web-based interventions (Boß et. al 2016) and has been used in previous studies to evaluate satisfaction with mental health interventions (Bäuerle et. al 2021). Like the COMPI-FPSS, it utilizes a Likert scale. Participant scores will be added and analyzed for each question and overall. A higher score means higher satisfaction, while a lower score means less satisfaction.

The purpose of the survey completed immediately after enrollment is to collect demographic information and obtain baseline COMPI-FPSS scores. The surveys completed at the ten-week study time point (after the experimental group has completed the research-related intervention) will be used to evaluate any changes in COMPI-FPSS scores, to assess if other stress-reducing interventions outside of the study are being utilized by subjects, to assess adherence to the research-related intervention protocol, and to determine satisfaction with the research-related intervention and fertility treatment. The final survey, completed at the 16-week study time point, will be used to evaluate whether the OC method has a prolonged effect on stress levels (i.e., whether COMPI-FPSS scores are similar to scores at week 10), to assess if other stress-reducing interventions outside of the study are being utilized by subjects, to assess continued interaction with the study materials after completion of the ten-week research-related intervention, and to explore continued satisfaction with the research-related intervention and fertility treatment (i.e., whether the perception of the research-related intervention remains the same).

Following completion of the first survey, participants randomized to the control group will receive standard fertility care, which does not currently include any stress-decreasing interventions or information. The control group will have access to the OC materials after the study period. Participants in the intervention group will begin the OC research-related intervention that will last ten weeks. Participants' fertility journey will not be delayed while they complete the intervention. Rather, it will happen simultaneously. The study team will be collaborating with OC who designed a ten-week curriculum that includes all the materials their clients already engage with. The curriculum will involve assignments that will take approximately three hours per week to complete and biweekly support group sessions with a certified coach. Participants will also have the option to join the Organic Conceptions Facebook group. The group sessions will be attended by both subjects and OC clients. Before every group call, participants will be sent a reminder message with instructions on how to remain anonymous during the sessions, if they wish to do so. To verify that participants are completing modules, the OC portal has the ability to track their completion. In addition, subjects will be asked the extent to which they are interacting with the assignments, how many support group sessions they attended, and whether they joined the Facebook group as part of their surveys. However, they will not be asked to turn in their workbook due to their private nature.

To evaluate whether providing the OC research-related intervention increases the subject's likelihood of attending their initial appointment, completing the fertility testing and treatment process, patient retention, conversion, and completion rates will be measured. Subjects will be considered "retained" if they attend their initial appointment and return for their follow-up appointment within six months of their initial consultation. If they do not return or return later than 6 months, they will be considered "unretained." Similarly, subjects will be considered "converted" if they enter a fertility treatment cycle within six months of their follow-up visit. If they do not, they will be considered "unconverted." Subjects will be considered "complete" if they complete their fertility treatment cycle. If they do not, they will be considered "incomplete." In addition, study participants will be asked whether they conceived (experienced a positive pregnancy test, confirmed by blood work) as part of the surveys completed at the ten-week and 16-week time points in the study. The electronic medical record system will be used to verify this information. If they do not conceive during the study period, their charts will continue to be monitored in the medical record system for one year.

ELIGIBILITY:
Inclusion Criteria:

* Speaks and reads English
* New patient at Shady Grove Fertility in Roanoke or Richmond
* Access to smartphone, tablet, or computer, and internet

Exclusion Criteria:

* Has seen a fertility specialist (reproductive endocrinologist) before AND underwent fertility treatment under that provider
* Is currently engaging with the Organic Conceptions method

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Stress levels in women with infertility | Day 0, end of week 10 (day 70), end of week 16 (day 112)
  Measured by responses to the Copenhagen Multi-center Psychosocial Infertility Fertility Problem Stress Scale Minimum value: 14 Maximum value: 66 Higher score means higher stress level due to infertility, and a potentially worse outcome

SECONDARY OUTCOMES:
Comparison of number of participants in each study group who returned for follow-up appointment within 6 months of initial consultation | Within 6 months of initial consultation
  Returning for follow-up appointment
Comparison of number of participants in each study group who began fertility treatment within 6 months of follow-up appointment | Within 6 months of follow-up appointment
  Beginning fertility treatment
Comparison of number of participants in each study group who completed fertility treatment | Recorded immediately after fertility treatment (IVF, ovulation induction, etc) is completed. Depends upon the treatment and what the provider indicates the treatment path should be
  Completed fertility treatment
Pregnancy rates | Study period (16 weeks) + 1 year
  Pregnancy outcome measured in three surveys and through monitoring of EMR
Satisfaction with Organic Conceptions intervention | End of week 10 (day 70), end of week 16 (day 112). Intervention group only.
  Measured by responses to Client Satisfaction Questionnaire for Internet Interventions Minimum value: 8 Maximum value: 32 Higher score means higher satisfaction with Organic Conceptions intervention.
Satisfaction with treatment | End of week 10 (day 70), end of week 16 (day 112)
  Measured by responses to survey questions (Likert scale) Minimum value = 1 Maximum value = 5 Higher score means higher satisfaction with fertility treatment.
Longevity of the effect of the intervention | End of week 10 (day 70), end of week 16 (day 112)
  Measured by comparing responses to the Copenhagen Multi-center Psychosocial Infertility Fertility Problem Stress Scale from the second and third survey. If score decreased from first to second survey, and score was similar/greater on third survey, then intervention has a long-lasting effect on stress levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Shady Grove Fertility, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No